CLINICAL TRIAL: NCT03202524
Title: Fresh Frozen Plasma as a Substitute for Albumin in Patients Receiving a Large Volume Paracentesis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was never approved by the IRB
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-8009
Record Dates: First submitted 2017-06-08; First posted 2017-06-28 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Liver Cirrhosis; Ascites Hepatic
Keywords: Paracentesis; Albumin; Plasma
MeSH Terms: conditions — Liver Cirrhosis | interventions — Albumins

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Albumin (Active Comparator): Patients undergoing large volume paracentesis with receive 50ml of 25% albumin for every 2 L removed from their abdomen.
  Interventions: Biological: Albumin
- Fresh Frozen Plasma (Experimental): Patients undergoing large volume paracentesis with receive 2 units of FFP for the first 4L removed followed by 50ml of 25% albumin for every additional 2 L removed
  Interventions: Biological: Fresh Frozen Plasma (FFP)

INTERVENTIONS:
Biological: Fresh Frozen Plasma (FFP) — FFP will be used as a substitute for albumin for the prevention of post-paracentesis circulatory dysfunction.
  Arms: Fresh Frozen Plasma
Biological: Albumin — Albumin will be used for the prevention of post-paracentesis circulatory dysfunction, as is the standard of care
  Arms: Albumin

SUMMARY:
Large volume paracentesis with albumin administration is the standard of care for patients with refractory ascites complicating end-stage liver disease. However, the use of albumin is frequently limited due to expense and occasional short supply. The goal of this study is to demonstrate if the administration of fresh frozen plasma (FFP) is as effective as albumin for volume expansion at the time of a large volume paracentesis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Cirrhosis of the liver based on biopsy or clinical and radiographic criteria
3. Ability to provide informed consent (Grade 0 to 1 HE)
4. Grade 3 ascites or refractory ascites
5. Ascites requiring frequent large volume paracentesis of at least 5 liters at least once a month
6. No diuretic use

Exclusion Criteria:

1. Inability to obtain informed consent
2. Age less than 18
3. Hepatic Encephalopathy Grade > 1
4. Septic shock
5. Active infection
6. Respiratory failure
7. Heart failure with reduced ejection fraction of ≤ 50%
8. Moderate or severe pulmonary hypertension
9. History of stroke
10. Unstable coronary artery disease
11. Chronic kidney disease (GFR <60)
12. GI bleed within 2 weeks
13. Any licorice within 2 weeks of starting the study
14. Any Beta Blocker use within the last 2 weeks
15. Any diuretic use within 2 weeks
16. Absence of paracentesis within 2 weeks
17. Absence of volume expanders within 2 weeks
18. INR > 1.7

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of Post-Paracentesis Circulatory Dysfunction (PPCD) | 6 Days
  The development of PPCD is diagnosed by an increase in plasma renin activity of more than 50% of baseline to > 4 ng/mL/h on the 6th day post paracentesis

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Sigal, MD, Principal Investigator — Montefiore Medical Center

IPD SHARING:
Plan to Share IPD: No
Data collected during the study will only be shared with researchers approved to key-personnel on the study protocol.